CLINICAL TRIAL: NCT04051359
Title: Effectiveness and Safety of Two Different Diets in Terms of Carbohydrate Restriction in Pregnant Women With Gestation Diabetes Mellitus
Brief Title: Carbohydrate Restriction in Pregnant Women With Gestation Diabetes Mellitus
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Tel-Aviv Sourasky Medical Center (Other Government)
Responsible Party: Principal Investigator, michal roll, PA, Tel-Aviv Sourasky Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 0244-18-TLV
Record Dates: First submitted 2019-08-08; First posted 2019-08-09 (Actual); Last update posted 2019-08-09 (Actual); Status verified 2019-08

CONDITIONS: Gestational Diabetes
MeSH Terms: conditions — Diabetes, Gestational | interventions — Diet

STUDY DESIGN:
Intervention Model Description: Randomized trial
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Standard carbohydrate (200 g) group (Active Comparator): Assignment to treatment groups will be performed on the enrollment to the study by evaluating the dietary carbohydrate intake personal patient preferences from 3 days prospective 24 hours' food dairy. After, the randomization will be performed and GDM patients will be assigned to the standard carbohydrate (200 g) group.
  Interventions: Other: Low carbohydrate (130 g) diet
- Low carbohydrate (130 g) group (Experimental): Assignment to treatment groups will be performed on the enrollment to the study by evaluating the dietary carbohydrate intake personal patient preferences from 3 days prospective 24 hours' food dairy. After, the randomization will be performed and GDM patients will be assigned to the low carbohydrate (130 g) group.
  Interventions: Other: Low carbohydrate (130 g) diet

INTERVENTIONS:
Other: Low carbohydrate (130 g) diet — Isocaloric moderately reduced carbohydrate diet (RCD, reduced carbohydrate diet) (~130 grams of carbohydrates)

SUMMARY:
The purpose of this controlled, randomized intervention is to investigate whether a carbohydrate-restricted diet, having a positive effect on blood sugar and weigh maintaining in diabetes, is effective and safe for pregnant woman with GDM and safe for their offspring, when compared to the standard carbohydrate content diet.

DETAILED DESCRIPTION:
Increasing prevalence of obesity and tendency to become pregnant later in life can explain rising prevalence of gestation diabetes (GDM) (1). Diabetes in pregnancy is a major public health issue: it has been shown that the mother's glycemic levels correlates perfectly with child's birth weight, death in utero, perinatal mortality and hypoglycemia (2). Therapeutic management is relatively simple and based on correction of hyperglycemia by carbohydrate restriction and energy-controlled diet adapted to pre-pregnancy BMI (3).

Although restriction of dietary carbohydrate has been the cornstone for treatment of GDM (4,5) with ACOG and The Endocrine Society recommendation for carbohydrate intake to 33-40% of total daily calories, the paucity of RCT evidence supporting safety of carbohydrate restriction still exist and actual dietary composition that optimizes perinatal outcomes is unknown (3).

Carbohydrate restriction in GDM comes with the potential increases in dietary fat intake and consequently a strong association between maternal lipids (i.e., triglycerides and free fatty acids) and excess fetal growth (6). Moreover, restrictive caloric and carbohydrate diet increases ketogenesis and ketone bodies (acetoacetate and beta-hydroxybutyrate (BHB) cross well the placental barrier.

Gestational ketogenic diet in mouse deleteriously affects the offspring growth and brain development (7), an early postnatal exposure to a ketogenic diet results in significant alterations to neonatal brain structure and can be accompanied by functional and behavioral changes in later postnatal life (8).

In the second half of pregnancy, under the influence of increasing placental hormones and cytokine concentration, lipolysis become dominant and use of free fatty acids as the energy material for the mother's body in place of glucose that is consumed mostly by the fetus.

These mechanisms are responsible for increased ketogenesis during pregnancy and are three times higher at night among pregnant women than among nonpregnant women (16). Human studies focused mostly exclusively on ketonuria; and a negative correlation between ketonuria and intellectual quotient in children born to diabetic mothers have been reported (9). Rizzo et al. did not confirm this correlation, although the authors did reveal a negative correlation between maternal β-hydroxybutyrate concentration in blood and the child's mental development (10).

On the other hand, evaluating ketone production in early pregnancy with type 1 diabetes by measuring blood BHB, the Jovanovic et al. found that despite the significantly elevated blood BHB level (2.5-fold higher than nondiabetic pregnant at 6th week gestation, and 1.6-fold at 12th week gestation), there was trend to lower BHB level in diabetic and nondiabetic mothers with malformed infants and pregnancy loss. The level of BHB was lower also in diabetic mothers of macrosomic infants (11).

Recently, inexpensive quantitative test of BHB became available using small capillary blood sample. Therefore, we would like to evaluate the levels of BHB in GDM patients treated by two different carbohydrate restricted diets in order to add an evidence on safety and proper caloric and carbohydrate restriction recommendation during pregnancy in order to optimize maternal and perinatal outcomes.

ELIGIBILITY:
Inclusion Criteria:

1. Ages 18-45 years
2. GDM diagnosed between 12 and 34 weeks gestation according to Carpenter and Coustan criteria (13)
3. BMI 20-35 kg/m2
4. Singleton pregnancy
5. Willing to perform self-monitoring of blood glucose at least 4 times a day
6. Self-monitoring of blood glucose
7. 12 to 34 weeks of gestation at the time of randomization
8. Signed informed consent

Exclusion Criteria:

1. Pre-existing diabetes in pregnancy, including first trimester fasting glucose ≥105 mg/dL
2. Use of other oral hypoglycemic agents during this pregnancy
3. Multiple pregnancy
4. Known hepatic insufficiency (bilirubin >50 µmol/L and/or protrombin time <50 %)
5. Insufficient understanding
6. Participant in another investigational drug study at inclusion visits
7. Fetal malformation diagnosed by previous fetal ultrasound

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 110 (Estimated)
Dates: Start 2019-08-15 (Estimated); Primary Completion 2021-02-15 (Estimated); Study Completion 2021-08-15 (Estimated)

PRIMARY OUTCOMES:
The rate of treatment failure defined as patients needing additional hypoglycemic therapy by long-insulin acting analogue detemir evaluated by capillary glucose levels | From one week after inclusion : 13 to 36 weeks of gestation to delivery
  o The treatment failure would be defined if the fasting SMBG would be ≥95 mg/dl and/or if 1-hour post-prandial (PP) BG would be ≥140 mg/dl or 2 hour PP BG would be ≥120 mg/dl in >20% of the measurements

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Endocrinology, Metabolism and Hypertension, Tel-Aviv Sourasky Medical Center, Tel Aviv, Israel

IPD SHARING:
Plan to Share IPD: Undecided
All women will be instructed to keep a diet of 25 kcal/kg/day for overweight and obese (pre-pregnancy BMI >25) and 35 kcal/kg for women with normal weight (pre-pregnancy BMI 18.5-24.9).
  The intervention (low carbohydrate intake = RCD) group will be instructed to keep a diet divided into 3 full meals and four snacks of 130 g/d (or at least 20% of total daily caloric intake) of carbohydrate intake and high protein and high fat intake from plant-source foods (35-55% fat, and 20-25% protein). Protein content will be the same amount in both groups.
  The standard carbohydrate diet (control group) group will be instructed to keep a diet divided into 3 full meals and four snacks of 200 g/d (or at least 40% of total daily caloric intake) of carbohydrate intake and high protein and high fat intake from plant-source foods (35-45% fat, and 20-25% protein).